CLINICAL TRIAL: NCT00548977
Title: Genetic Studies Spermatogenic Failure
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Other Study IDs: NCKUH-1
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Last update posted 2007-10-25 (Estimated); Status verified 2007-10

CONDITIONS: Oligospermia; Azoospermia; Male Infertility
Keywords: spermatogenesis defect; male infertility; azoospermia; oligozoospermia; Y chromosome markers; estrogen gene
MeSH Terms: conditions — Oligospermia; Azoospermia; Infertility, Male

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Drawing blood to study genetic polymorphism

SUMMARY:
The proposed study is designed to test the following hypotheses:

1. Mouse autosomal or X-linked genes which are exclusively expressed in mouse spermatogonia are also spermatogonia-specific in human.
2. Severe spermatogenic defect, especially hypospermatogenesis or SCOS, is caused by an intrinsic defect in germ line stem cell or speramtogenia.
3. Spermatogonia-specific genes are caudate genes for human spermatogenic defect, especially for hypospermatogenesis or SCOS.
4. For a significant fraction of cases with severe spermatogenic defect, the sterile genes are transmitted via multifactorial inheritance mode.
5. For some cases with severe spermatogenic defect, mutations of spermatogonia- specific genes may be transmitted in the X-linked recessive, autosomal recessive, or autosomal dominant mode.

DETAILED DESCRIPTION:
Between 2% and 12% of couples worldwide are affected by reduced fertility. Men who have defects in sperm production (spermatogenic defect) account for about half of these cases. In Drosophila and mouse, targeted disruptions of numerous sterility- associated genes have been created. Physiological studies in the Drosophila and in mouse also indicate that spermatogenesis is subjected to complex regulation, and male infertility may result from aberrant regulatory events. In the human being, deletions of the Y chromosome account for only 10% of cases with spermatogenic defect, and etiologies of remaining 90% of cases are still unknown. It is evident that multiple genes are involved in male infertility. For cases with severe spermatogenic defect , testicular histology shows either decreased number of germ cells in all developmental stages (hypospermatogenesis) or complete absence of germ cells (Sertoli cell only syndrome or SCOS). It appears that there is an intrinsic defect which causes depletion of germ-line stem cells (spermatogonia) for cases with hypospermatogenesis or SCOS. Of 25 genes exclusively expressed in mouse spermatogonia, 3 are Y-linked, 10 are X-linked, and only 12 are distributed on autosomes.

ELIGIBILITY:
Inclusion Criteria:

* Men with oligozoospermia(<2*10^7/ml) or azoospermia

Exclusion Criteria:

* Abnormal karyotypes
* Obvious genital trauma history
* Genital hernia
* Other recognizable causes of male infertility

Ages: 14 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patient visited our outpatient clinic
Sampling Method: Probability Sample
Enrollment: 283 (Actual)
Dates: Start 2001-01; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Genotype/phenotype correlation of Y-linked AZF candidates and estrogen-related genes | At the time of visiting OPD

SECONDARY OUTCOMES:
Role of significant candidate genes in human spermatogenesis | At the time of drawing blood

CONTACTS AND LOCATIONS:
Overall Officials: Paolin Kuo, MD, Study Chair
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan